CLINICAL TRIAL: NCT03456830
Title: Evaluate the Safety and Efficacy of ALLN-177 in Patients With Enteric Hyperoxaluria: A Phase III Randomized, Placebo-Controlled Study
Brief Title: Evaluate ALLN-177 in Patients With Enteric Hyperoxaluria
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allena Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALLN-177-301
Record Dates: First submitted 2018-03-01; First posted 2018-03-07 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: Enteric Hyperoxaluria
Keywords: Kidney stones; Hyperoxaluria; Enteric hyperoxaluria; Oxalate
MeSH Terms: conditions — Kidney Calculi; Hyperoxaluria | interventions — reloxaliase; oxalate decarboxylase

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ALLN-177 (Experimental): ALLN-177 3,750 units per capsule
  Interventions: Drug: ALLN-177
- Placebo (Placebo Comparator): Placebo capsule
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALLN-177 — ALLN-177 7,500 units (2 capsules), orally, with each meal/snack, 3 to 5 times per day for 28 days
  Other Names: Oxalate decarboxylase
  Arms: ALLN-177
Drug: Placebo — Placebo 2 capsules, orally, with each meal/snack, 3 to 5 times per day for 28 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the efficacy and safety of ALLN-177 in patients with enteric hyperoxaluria.

DETAILED DESCRIPTION:
This is a phase 3, multicenter, randomized, double-blind, placebo-controlled study. This study is designed to determine whether treatment with ALLN-177 for 28 days can reduce urinary oxalate excretion in patients with enteric hyperoxaluria and to evaluate the safety of ALLN-177 in this patient population compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Provided informed consent
2. Age 18 or older
3. History of hyperoxaluria secondary to a known underlying enteric disorder associated with malabsorption (e.g., bariatric surgery, Crohn's disease, short bowel syndrome, or other malabsorption syndrome)
4. Urinary Oxalate ≥ 50mg/24h

Exclusion Criteria:

1. Acute renal failure or estimated glomerular filtration rate (eGFR) < 30mL/min/1.73 m2
2. Unable or unwilling to discontinue Vitamin C supplementation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-10-28 (Actual)

PRIMARY OUTCOMES:
Percent change from baseline in 24-hour urinary oxalate excretion during Weeks 1-4 | 4 weeks
  Efficacy will be assessed based on percent change from baseline to the mean of Weeks 1-4, derived from all 24-hour collections during Weeks 1-4 on treatment

SECONDARY OUTCOMES:
Proportion of subjects with a ≥ 20% reduction from Baseline in 24-hour urinary oxalate excretion during Weeks 1-4 | 4 weeks
  Efficacy will be assessed based on proportion of subjects with ≥ 20% reduction from baseline to the mean of Weeks 1-4, derived from all 24-hour collections during Weeks 1-4 on treatment

CONTACTS AND LOCATIONS:
Overall Officials: Annamaria Kausz, MD MS, Study Director — Allena Pharmaceuticals Inc
Locations (63):
- United States (39):
  - Urology Centers of Alabama, Birmingham, Alabama
  - University of Alabama, Department of Urology, Birmingham, Alabama
  - Mayo Clinic Hospital, Phoenix, Arizona
  - Urological Associates of Southern Arizona, Tucson, Arizona
  - Applied Research Center of Arkansas, Little Rock, Arkansas
  - TROVARE Clinical Research, Bakersfield, California
  - Advanced Urology Institute, Daytona Beach, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Center for Advanced GI (CFAGI), Maitland, Florida
  - South Medical Research Group, Inc., Miami, Florida
  - North Idaho Urology, Coeur d'Alene, Idaho
  - Idaho Urologic Institue, Meridian, Idaho
  - Edmund J. Lewis and Associates, Chicago, Illinois
  - IU Health Physicians, Indianapolis, Indiana
  - Regional Urology, Shreveport, Louisiana
  - Maine Nephrology Associates, Portland, Maine
  - Pen Bay Medical Center, Rockport, Maine
  - Chesapeake Urology, Hanover, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mayo Clinic-Dept. of Nephrology, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - The Urology Center, P.C., Omaha, Nebraska
  - Park Avenue Endocrinology & Nutrition, New York, New York
  - Columbia University Medical Center, New York, New York
  - Advanced Urology Centers of New York, Plainview, New York
  - Albert Einstein College of Medicine Montefiore Medical Center, The Bronx, New York
  - University of North Carolina Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Associated Urologists of North Carolina, Raleigh, North Carolina
  - Coastal Urology, Wilmington, North Carolina
  - Tristate Urologic Services PSI Inc, Cincinnati, Ohio
  - Genito-Urinary Surgeons, Toledo, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Houston Nephrology Group, Cypress, Texas
  - Renal Disease Research Institute, Dallas, Texas
  - Houston Metro Urology, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Virginia Urology, Richmond, Virginia
  - Urology of Virginia, Virginia Beach, Virginia
- Canada (5):
  - University of Alberta, Division of Urology, Edmonton, Alberta
  - Silverado Research Inc, Victoria, British Columbia
  - Toronto Digestive Disease Associates, Inc., Vaughan, Ontario
  - Centre de Recherche du Centre Hospitalier de l'Université de Montréal (CRCHUM), Montreal, Quebec
  - Research center of CHU de Québec - Université Laval (CHUL), Québec, Quebec
- CHU de Nancy-Hopital Brabois, Vandœuvre-lès-Nancy, France
- Germany (7):
  - Charite Universitaetsmedizin Berlin, Berlin
  - Universitat Bonn - Zentrum für Kinderheilkunde, Bonn
  - Universitaetsklinikum Bonn; Klinik und Poliklinik für Urologie und Kinderurologie, Bonn
  - Universitatsklinikum Freiburg, Klinik for Urologie, Freiburg im Breisgau
  - Universitaetsklinikum Leipzig, Leipzig
  - PSHI GmbH; PFÜTZNER Science & Health Institute GmbH, Mainz
  - Universitat Munchen - Großhadern, Munich
- Italy (4):
  - IRCCS Azienda Ospedaliera Universitaria San Martino IST, Genova
  - ASST di Lecco, Lecco
  - Azienda Socio-Sanitaria Territoriale di Lecco (ASST di Lecco), Lecco
  - Fondazione Policlinico Universitario A. Gemelli - Universita Cattolica del Sacro Cuore, Rome
- Spain (5):
  - Hospital Universitari de Girona Doctor Josep Trueta, Girona
  - Complejo Asistencial de León, León
  - Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario Infanta Sofia, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
- United Kingdom (2):
  - The Royal Free Hospital, London
  - Freeman Hospital, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Langman CB, Grujic D, Pease RM, Easter L, Nezzer J, Margolin A, Brettman L. A Double-Blind, Placebo Controlled, Randomized Phase 1 Cross-Over Study with ALLN-177, an Orally Administered Oxalate Degrading Enzyme. Am J Nephrol. 2016;44(2):150-8. doi: 10.1159/000448766. Epub 2016 Aug 17. PMID 27529510
- [Derived] Lieske JC, Lingeman JE, Ferraro PM, Wyatt CM, Tosone C, Kausz AT, Knauf F. Randomized Placebo-Controlled Trial of Reloxaliase in Enteric Hyperoxaluria. NEJM Evid. 2022 Jul;1(7):EVIDoa2100053. doi: 10.1056/EVIDoa2100053. Epub 2022 May 6. PMID 38319254